CLINICAL TRIAL: NCT00000638
Title: Prophylaxis Against Tuberculosis (TB) in Patients With Human Immunodeficiency Virus (HIV) Infection and Confirmed Latent Tuberculous Infection
Brief Title: Preventive Treatment Against Tuberculosis (TB) in Patients With Human Immunodeficiency Virus (HIV) Infection and Confirmed Latent Tuberculous Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoechst Marion Roussel (Industry); Lederle Laboratories (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: ACTG 177; CPCRA 004; TB/PPD+; 11152 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; Isoniazid; Mycobacterium tuberculosis; Pyrazinamide; Pyridoxine; Rifampin; AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antitubercular Agents; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Tuberculosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Isoniazid; Pyrazinamide; Pyridoxine; Rifampin

INTERVENTIONS:
Drug: Isoniazid
Drug: Pyrazinamide
Drug: Pyridoxine hydrochloride
Drug: Rifampin

SUMMARY:
To evaluate and compare the safety and effectiveness of a one-year course of isoniazid (INH) versus a two-month course of rifampin plus pyrazinamide for the prevention of reactivation tuberculosis in individuals infected with both HIV and latent (inactive) Mycobacterium tuberculosis.

Current guidelines from the American Thoracic Society and the Centers for Disease Control recommend 6 to 12 months of INH for PPD (purified protein derivative)-positive individuals. Although the effectiveness of this treatment is not known for HIV-infected individuals, several studies using INH to prevent tuberculosis in presumably normal hosts have shown 60 to 80 percent effectiveness. Problems with this treatment include compliance, adverse reaction, and the possibility of not preventing disease due to tuberculosis organisms being resistant to INH. A two-month preventive treatment plan should help in increasing compliance. In addition, the use of two drugs (rifampin / pyrazinamide) may help overcome problems with drug resistance. If this study shows equal or greater effectiveness of the two-month rifampin / pyrazinamide treatment, it could alter the approach to tuberculosis prevention for both HIV-positive and HIV-negative individuals.

DETAILED DESCRIPTION:
Current guidelines from the American Thoracic Society and the Centers for Disease Control recommend 6 to 12 months of INH for PPD (purified protein derivative)-positive individuals. Although the effectiveness of this treatment is not known for HIV-infected individuals, several studies using INH to prevent tuberculosis in presumably normal hosts have shown 60 to 80 percent effectiveness. Problems with this treatment include compliance, adverse reaction, and the possibility of not preventing disease due to tuberculosis organisms being resistant to INH. A two-month preventive treatment plan should help in increasing compliance. In addition, the use of two drugs (rifampin / pyrazinamide) may help overcome problems with drug resistance. If this study shows equal or greater effectiveness of the two-month rifampin / pyrazinamide treatment, it could alter the approach to tuberculosis prevention for both HIV-positive and HIV-negative individuals.

Patients are chosen by a random selection process to either the INH or the rifampin / pyrazinamide arm of the dose. Patients on the INH arm receive INH plus vitamin B6 (pyridoxine hydrochloride ) daily for 12 months. Patients on the other arm receive rifampin plus pyrazinamide for 60 days. Dosage of rifampin and pyrazinamide depends on weight of patient.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral treatment.
* Pneumocystis carinii pneumonia prophylaxis.
* Treatment for acute opportunistic infection.

Patients must have:

* HIV infection.
* Current or documented history of positive PPD skin test.
* Life expectancy of at least 6 months or, in the physician's opinion, patient has a reasonable chance of survival to end of study.

Allowed:

* Participation in other clinical trials as long as there is no potential activity of other study drugs against Mycobacterium tuberculosis (MTb), additive toxicities between study agents, or known possible drug interactions between study drugs.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Current active clinical tuberculosis, confirmed or suspected.
* History of sensitivity / intolerance to any study medication.
* Evidence of peripheral neuropathy, i.e., signs or symptoms of paresis, paresthesias, neuromotor abnormalities, or neurosensory deficits of grade 3 or worse.
* Unwilling or unable to have current therapy and/or concomitant medication changed to avoid serious interaction with study medication.
* Acute hepatitis.
* Unable to comply with the follow-up requirements of the protocol.

Concurrent Medication:

Excluded:

* Treatment with quinolones, fluoroquinolones, aminoglycosides, or other agents that have activity against Mycobacterium tuberculosis.
* Excluded as ongoing (i.e., continuous, chronic and/or recurring) treatment:
* Aminoglycosides such as amikacin, aminosalicylic acid salts (PAS), capreomycin, clofazimine, cycloserine, ethambutol, ethionamide, isoniazid (INH) if randomized to rifampin/pyrazinamide arm of study, kanamycin, pyrazinamide if randomized to INH arm of study, and quinolones and fluoroquinolones, i.e., rifabutin, rifampin (if randomized to INH arm of study), ciprofloxacin, levofloxacin, ofloxacin, streptomycin, and thiacetazone.

Prior Medication:

Excluded:

* More than 2 months of continuous treatment, after documentation of a positive PPD skin test, with agents that have known or potential antituberculous activity or any antimycobacterial medication for > 1 month.

Patients may not have the following prior conditions:

* History of sensitivity / intolerance to any study medication.
* Unwilling or unable to comply with the follow-up requirements of the protocol.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Study Completion 1999-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaisson R, Study Chair
Locations (76):
- United States (75):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hosp of Los Angeles, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Olive View Med Ctr, Sylmar, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Yale Univ / New Haven, New Haven, Connecticut
  - HIV Ctr - District of Columbia Gen Hosp, Washington D.C., District of Columbia
  - Whitman - Walker Clinic / Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Children's Mem Hosp Family Cln / Northwestern Univ Med Schl, Chicago, Illinois
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Adirondack Med Ctr at Saranac Lake, Albany, New York
  - Albany Med College / Division of HIV Medicine A158, Albany, New York
  - Mid - Hudson Care Ctr, Albany, New York
  - Interfaith Med Ctr, Brooklyn, New York
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Nassau County Med Ctr, East Meadow, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - North Shore Univ Hosp, Manhasset, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Comprehensive Health Care Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Samaritan Village Inc / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Wake County Dept of Health, Raleigh, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Girard Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Med Univ of South Carolina / UNC, Charleston, South Carolina
  - Julio Arroyo, West Columbia, South Carolina
  - Meharry Med College, Nashville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Houston Clinical Research Network, Houston, Texas
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Halsey N, et al. Twice weekly INH vs RIF and PZA for TB prophylaxis in HIV infected adults. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:55
- [Background] Gordin F, Chaisson RE, Matts JP, Miller C, de Lourdes Garcia M, Hafner R, Valdespino JL, Coberly J, Schechter M, Klukowicz AJ, Barry MA, O'Brien RJ. Rifampin and pyrazinamide vs isoniazid for prevention of tuberculosis in HIV-infected persons: an international randomized trial. Terry Beirn Community Programs for Clinical Research on AIDS, the Adult AIDS Clinical Trials Group, the Pan American Health Organization, and the Centers for Disease Control and Prevention Study Group. JAMA. 2000 Mar 15;283(11):1445-50. doi: 10.1001/jama.283.11.1445. PMID 10732934